CLINICAL TRIAL: NCT04450095
Title: Effects of Endothelin Receptor Antagonist on Ischemic Kidney Injury During Nephron Sparing Surgery for Renal Mass Excision: Assessment by Ischemia Biomarkers, NGAL, KIM-1
Brief Title: Effects of Endothelin Receptor Antagonist on Ischemic Kidney Injury During Nephron Sparing Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ofir. Avitan, Dr. Avitan Ofir, Bnai Zion Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 0048-18-BNZ
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Kidney Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated group (Active Comparator): Tab. Volibris 10mg given once a day for 5 days, starting 48 hours before surgery (in addition for the standard treatment for partial nephrectomy)
  Interventions: Drug: Ambrisentan 10 MG
- Control group (No Intervention): Treated with the standard treatment for partial nephrectomy

INTERVENTIONS:
Drug: Ambrisentan 10 MG — be given once a day for 5 days, starting 48 hours before surgery
  Arms: Treated group

SUMMARY:
Based on animal studies, it was found that administration of endothelial receptor antagonists before and after renal blood vessels clamp and release results in a significantly reduced renal function injury.

On the basis of these results, we chose to divide the study population into 2 groups: control group that would be treated the standard accepted preventive treatment: intravenous injection of Mannitol, cooling of the kidney surface, compared to the treatment group that in addition would receive pre- and post-operative treatment of endothelial receptor antagonists (Ambrisentan (Volibris (10mg).

To be noticed that the drug is recognized and is given as a primary indication for patients with pulmonary hypertension.

The differences between the renal function and biomarkers for pre- and post-operative renal ischemic injury would be examined in order to disclose if the kidney injury of the treated group was indeed smaller.

This information will enable us to protect the operated kidneys from the ischemic damage, especially in those patients with poor basic renal function.

DETAILED DESCRIPTION:
This is a study aimed at examining the protective effect of endothelin antagonism on the ischemic damage the kidney undergoes during partial nephrectomy for kidney lesion removal.

In such procedure, it is common to clamp the kidney blood vessels in order to eliminate blood flow in the surgical field that will enable clear visibility to differentiate the tumor tissue from the normally kidney parenchyma.

Later, after removing the tumor lesion and suturing the tumor bed, the blockage is released and the renal blood flow returns.

The blockage itself and its release causes damage to the kidney tissue that is usually reduced by the kidney's cooling (through ice crystals)and as well as intravenous injection of mannitol.

In this study, patients were divided into 2 groups randomly, assigned the receipt in the order of recruitment.

The first group will receive the standard treatment and the other will be given before and after surgery endothelin antagonists in addition to the standard treatment. The drug will be given once a day for 5 days, starting 48 hours before surgery. Treatment efficacy assessment will be based on comparison of renal function (serum creatinine level and glomerular filtration) as well as biomarkers of acute renal damage (NGAL, KIM-1, and others) that will be taken from patients before and at different time points after surgery: urine samples to be taken at the following time points: - 3 , 8,24,48,72 hours after surgery. Blood samples will be taken at the following time points: - 8, 24, 48, 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a single kidney lesion who undergo Contrast enhancement (by CT scan)
2. Normal contra-lateral kidney as illustrated by imaging tests
3. Patients eligible for anesthesia and surgery

Exclusion Criteria:

1. Patients with chronic kidney infections
2. Blood clot disorders
3. End-stage renal failure
4. Patients sensitive to the study drug
5. Patients with cardiac heart failure, EF <40%
6. Patients with hyperkalemia
7. Patients with systolic blood pressure under 90 mmHg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
RENAL FUNCTION INJURY | 2 YEARS
  quantified by serum CRE, KIM-1,NGAL and urine markers KIM-1 NGAL

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Avitan, M.D., Principal Investigator — Bnai-zion medical center, Haifa, Israel
Locations (2):
- Israel (2):
  - Bnai-Zion Medical Center, Haifa
  - Department of Physiology, The Bruce and Ruth Rapapport Faculty of Medicine, Technion, Haifa

IPD SHARING:
Plan to Share IPD: No
Only the Patients index and the collected data will be provided without private names or ID numbers